CLINICAL TRIAL: NCT07172230
Title: Immersive Virtual Reality Induces Procedural Analgesia, Anxiolysis and Anterograde Amnesia: A Randomized Controlled Study 1
Brief Title: The Effective of Immersive Virtual Reality Distraction on Memory: Study 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Hunter Hoffman, Director, Virtual Reality Research Center at the Human Photonics Lab; Research Scientist:Dept of Mechanical Engineering, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: VRAnalgesia2025a
Record Dates: First submitted 2025-09-03; First posted 2025-09-15 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Healthy Participants
Keywords: Virtual reality amnesia

STUDY DESIGN:
Intervention Model Description: One within-subject randomized studies will be conducted in healthy adults. In Study 1 (n=16), participants will complete immediate free recall after hearing a 15-word list during No VR versus during immersive VR.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immersive virtual reality (Experimental): VR
  Interventions: Behavioral: Immersive Virtual Reality
- No VR (Other): No distraction during word list
  Interventions: Behavioral: No distraction Control condition

INTERVENTIONS:
Behavioral: Immersive Virtual Reality — Immersive VR
  Arms: Immersive virtual reality
Behavioral: No distraction Control condition — No VR during word list study phase
  Arms: No VR

SUMMARY:
The effect of virtual reality on memory.

DETAILED DESCRIPTION:
A within-subject randomized study will be conducted in healthy adults. In Study 1 (n=16), participants will complete immediate free recall after hearing a 15-word list during No VR versus during immersive VR.

ELIGIBILITY:
Inclusion Criteria:

* Currently enrolled in a course at the University of Washington Psychology Dept., participating in the University of Washington (UW) Psychology subject pool
* Able to read, write and comprehend English
* Able to complete study measures
* Willing to follow our UW approved instructions
* 18 years of age or older

Exclusion Criteria: People who have already previously participated in this same study (e.g., last quarter) are not eligible to participate again.

* Not enrolled in a course at the University of Washington Psychology Dept., not participating in the UW Psychology subject pool
* Not be able to read, write and comprehend English
* Younger than 18 years of age.
* Not capable of completing measures
* Not capable of indicating pain intensity,
* Not capable of filling out study measures,
* Extreme susceptibility to motion sickness,
* Seizure history,
* Unusual sensitivity or lack of sensitivity to pain,
* Sensitive skin,
* Sensitive feet
* Migraines
* Diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-05-31 (Actual); Primary Completion 2024-11-06 (Actual); Study Completion 2024-11-06 (Actual)

PRIMARY OUTCOMES:
Word Recall | begin 15 seconds after the last word
  Free immediate recall of each word study list, after each list
Distraction | Measured immediately after the free recall of word list 2
  Participants subjective ratings of how distracted they were in each condition

CONTACTS AND LOCATIONS:
Overall Officials: Hunter Hoffman, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
summarized aggregated data will be made available upon reasonable request
Time Frame: De-identified summarized aggregated data will be available upon publication in a peer reviewed journal until 2030
Access Criteria: summarized aggregate data will be made available upon reasonable request by e-mailing the primary contact.
URL: https://www.vrpain.com

REFERENCES:
- [Result] Hoffman HG, Fontenot MR, Garcia-Palacios A, Greenleaf WJ, Alhalabi W, Curatolo M, Flor H. Adding tactile feedback increases avatar ownership and makes virtual reality more effective at reducing pain in a randomized crossover study. Sci Rep. 2023 May 22;13(1):7915. doi: 10.1038/s41598-023-31038-4. PMID 37217536
- See also: website about VR analgesia — http://www.vrpain.com